CLINICAL TRIAL: NCT05985889
Title: Comparison of Innovative Rehabilitation Treatments and Examination of Their Effectiveness in Stroke Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Somogy Megyei Kaposi Mór Teaching Hospital (Other)
Responsible Party: Principal Investigator, Tollár József, Head of Department, Somogy Megyei Kaposi Mór Teaching Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IKEB/2023/01
Record Dates: First submitted 2023-08-02; First posted 2023-08-14 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Stroke
Keywords: robotic; stroke; rehabilitation; virtual rehabilitation
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Robotic (Experimental): They performed training with a robot 15 times over 3 weeks.
  Interventions: Other: Robot
- Fizio (Experimental): They receive physiotherapy treatment.
  Interventions: Other: Fizio
- EXE1 (Experimental): Virtual reality treatment is performed once a day.
  Interventions: Other: EXE1
- EXE2 (Experimental): Virtual reality treatment is performed twice a day.
  Interventions: Other: EXE2
- EXE+ROB (Experimental): Virtual and robotic treatments are performed once a day.
  Interventions: Other: EXE+ROB

INTERVENTIONS:
Other: Robot — You have to walk with a robot mounted on your lower limb. To move, to change direction.
  Other Names: ROB
  Arms: Robotic
Other: Fizio — Patients do state-funded physical therapy.
  Arms: Fizio
Other: EXE1 — Patients undergo intensive virtual reality therapy once a day.
  Arms: EXE1
Other: EXE2 — Patients undergo intensive virtual reality therapy twice a day.
  Arms: EXE2
Other: EXE+ROB — The patients intensively performed 1 virtual reality therapy and 1 robotic therapy every day.
  Arms: EXE+ROB

SUMMARY:
We perform a comparison of several groups. We would like to determine how robotic and virtual therapy is most effective in the treatment of stroke patients. We place great emphasis on walking speed, quality of life, coordination and changes in walking distance.

ELIGIBILITY:
Inclusion Criteria:

post stroke 6MWT : 120> minimum after stroke 3 days be a stroke patient first stroke hemiplegia

Exclusion Criteria:

multiple strokes, inability to stand and walk, cognitive function disorder does not reach 50 meters with a minimal walking aid Alcohol Sever heart problem sever demeanor alcoholism drug problems Drug

Ages: 55 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2023-07-08 (Actual); Primary Completion 2023-08-30 (Estimated); Study Completion 2023-08-30 (Estimated)

PRIMARY OUTCOMES:
mRS score | 3 weeks (0-5 score, high score better)

SECONDARY OUTCOMES:
Barthel index score | 3 weeks
Berg balance score | 3 weeks (0-30, high score better)
6MWT | 3 weeks
  meter
10m gait speed | 3 weeks
  m/s

CONTACTS AND LOCATIONS:
Locations (1):
- Dr. Tollár József, Kaposvár, Somogy County, Hungary

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/?term=soft+exosuit